CLINICAL TRIAL: NCT04837677
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation Study of PRT1419 in Patients With Advanced Solid Tumors
Brief Title: A Study of PRT1419 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT1419-02
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Sarcoma; Melanoma; Lung Cancer; Breast Cancer; Esophageal Cancer; Cervical Cancer; Head and Neck Cancer
Keywords: MCL1
MeSH Terms: conditions — Sarcoma; Melanoma; Lung Neoplasms; Breast Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT1419 (Experimental): PRT1419 will be administered by intravenous infusion
  Interventions: Drug: PRT1419

INTERVENTIONS:
Drug: PRT1419 — PRT1419 will be administered by intravenous infusion

SUMMARY:
This is a Phase 1 dose-escalation study of PRT1419, a myeloid cell leukemia 1 (MCL1) inhibitor, in patients with advanced solid tumors. The purpose of this study is to define the dosing schedule, maximally tolerated dose and/or estimate the optimal biological dose to be used in subsequent development of PRT1419.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation Phase 1 study of PRT1419, a MCL1 inhibitor, evaluating patients with relapsed or refractory solid tumors, including breast, lung, sarcoma and melanoma as part of a 28-day treatment cycle. The study will employ a "3+3" dose escalation design. The dose may be escalated until a dose limiting toxicity is identified.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Adequate organ function (bone marrow, hepatic, renal, cardiovascular)
* Left ventricular ejection fraction of ≥ 50%
* Female patients of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and must agree to use a highly effective method of contraception during the trial
* Patients must have recovered from the effects of any prior cancer related therapy, radiotherapy or surgery (toxicity ≤ Grade 1)
* All patients on prior investigational agents must wait at least 5 half-lives of the agent in question, or 28 days, whichever is longer before study entry
* Most recent lab values meet the following criteria:

  * Absolute neutrophil count > 1.0 x 10^3/μL;
  * Platelet count > 75,000/μL;
  * Hemoglobin > 9.0 g/dL
* Histologically confirmed advanced or metastatic solid tumor indicated below that is relapsed, refractory, or intolerant to available therapies with known benefit:

  * Sarcoma not amendable to curative treatment with surgery or radiotherapy;
  * Melanoma (non-resectable or metastatic);
  * Small cell lung cancer (extensive-stage);
  * Non-small cell lung cancer;
  * Triple negative breast cancer (histopathologically or cytologically confirmed).
  * Esophageal cancer
  * Cervical cancer
  * Head and neck cancer

Exclusion Criteria:

* Known hypersensitivity to any of the components of PRT1419
* Primary malignancies of the CNS, or uncontrolled CNS metastases, including impending spinal cord compression
* Female patients who are pregnant or lactating
* Inflammatory disorders of the gastrointestinal tract, or subjects with GI malabsorption
* Mean QTcF interval of >480 msec
* History of heart failure, additional risk factors for arrhythmias or requiring concomitant medications that prolong the QT/QTc interval
* HIV positive; known active hepatitis B or C
* Uncontrolled intercurrent illnesses
* Treatment with strong inhibitors of CYP2C8
* Prior exposure to an MCL1 inhibitor
* History of another malignancy except:

  * Malignancy treated with curative intent with no known active disease for >2 years at study entry;
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease;
  * Adequately treated carcinoma in situ without evidence of disease;
  * Other concurrent low-grade malignancies (i.e chronic lymphocytic leukemia (Rai 0)) may be considered after consultation with Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of PRT1419 | Baseline through Day 28
  Dose limiting toxicities will be evaluated through the first cycle
Maximally tolerated dose (MTD) and/or optimal biological dose (OBD) | Baseline through approximately 2 years
  The MTD and/or OBD will be established for further investigation in participants with advanced solid tumors.
Recommended phase 2 dose (RP2D) and schedule of PRT1419 | Baseline through approximately 2 years
  The RP2D will be established for further investigation in participants with advanced solid tumors.

SECONDARY OUTCOMES:
Safety and tolerability of PRT1419: AEs, SAEs, CTCAE assessments | Baseline through approximately 2 years
  Safety and tolerability will be assessed by recording adverse events (AEs) and serious adverse events (SAEs) according to Common Terminology Criteria for Adverse Events (CTCAE)
Pharmacokinetic profile of PRT1419: maximum observed plasma concentration | Baseline through approximately 2 years
  PRT1419 pharmacokinetics will be calculated including the maximum observed plasma concentration
Anti-tumor activity of PRT1419: measurement of objective responses | Baseline through approximately 2 years
  Anti-tumor activity of PRT1419 will be based on the measurement of objective responses
Progression-free survival | Baseline through approximately 2 years
  Progression-free survival will be calculated from the first administration of PRT1419 until death or until the criteria for disease progression are met

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Lake Mary, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee